CLINICAL TRIAL: NCT02688621
Title: Internet Assisted Obesity Treatment Enhanced With Financial Incentives
Acronym: iREACH3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: University of South Carolina (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jean R. Harvey, PhD, RD, Principal Investigator, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRBS 15-259; R01DK056746 (NIH)
Record Dates: First submitted 2016-02-09; First posted 2016-02-23 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Obesity
Keywords: weight loss; financial incentives; internet weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet only (Active Comparator): Participants will be required to attend a weekly Internet chat session with your group members and one of the behavioral weight control therapists. Participants will learn the principles of managing eating and exercise behaviors in weekly, hour-long chat sessions and by completing weekly lessons. Participants are asked to self-monitor foods and exercise through the use of a smartphone ap. Participants will wear a tracking device that monitors steps. All participants will be contacted via e-mail individually, by their group leader who will monitor their progress and offer advice and encouragement. Meetings are weekly for 24 weeks and monthly for 12 months.
  Interventions: Behavioral: Internet Only
- Internet + Incentives (Experimental): Participants are given the same intervention as described for the internet only group, with the exception that they will have the opportunity to earn financial incentives. Financial incentives will be based on participants weight loss, and compliance with certain weight loss behaviors including meeting exercise goals, self-monitoring foods consumed, and daily weighing and reporting.
  Interventions: Behavioral: Internet + Incentives

INTERVENTIONS:
Behavioral: Internet Only — 18 month behavioral weight loss intervention delivered online
  Arms: Internet only
Behavioral: Internet + Incentives — 18 month behavioral weight loss intervention delivered online with the possibility of earning incentives for losing weight and performing weight loss behaviors including monitoring food intake, exercising, and daily weighing
  Arms: Internet + Incentives

SUMMARY:
The investigators propose a randomized controlled trial to evaluate whether the addition of financial incentives to a high-quality, online behavioral weight loss intervention produces better weight losses than the online treatment alone.

DETAILED DESCRIPTION:
Overweight and obese but otherwise healthy participants (N=416) will be recruited in approximately equal numbers at two clinical centers, the University of South Carolina and the University of Vermont. Eligible participants will be randomized to one of two conditions: 1) an 18-month, 36-session group Internet behavioral weight control treatment (Internet Only) which replicates the intervention the investigators have implemented previously; or 2) the same 18-month, 36-session group Internet treatment plus financial incentives for performance of 3 key self-management behaviors (Internet+ Incentive). Both conditions will have access to the same web-based intervention platform and the same counselor-delivered intervention elements; the presence of economic incentives for behavioral and weight goals is the only difference between the conditions. Assessments will be conducted at Baseline, 2, 6, 12 and 18 months. Cost data will be collected to inform cost effectiveness evaluations.

ELIGIBILITY:
Inclusion Criteria:

* over 18
* BMI between 25 and 50
* Not currently pregnant or pregnant in the previous 6 months and currently breastfeeding or planning on becoming pregnant in 18 months
* Have a computer at home or at work with flashplayer, access to the internet, and a smart phone (to allow use of step counting aps)
* Free of medical problems that might contraindicate participation in a behavioral weight reduction program containing an exercise component
* Not enrolled in another weight reduction program
* Not currently on medication that would affect weight loss

Exclusion Criteria:

* had a heart attack or stroke in the previous six months
* had weight loss surgery
* lost 10 pounds or more in the previous 6 months
* currently taking medications for weight loss
* required by their doctor to follow a special diet (other than low fat)
* planning to move out of the area within 18 months
* schedule conflicts making it difficult to attend online "chats"
* live more than 60 minutes driving distance from either University of South Carolina or University of Vermont campuses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Delia Smith West, PhD, Principal Investigator — University of South Carolina; Jean R Harvey, PhD, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - University of South Carolina, Columbia, South Carolina
  - Behavioral Weight Management Program/Univ of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stansbury ML, Harvey J, Krukowski RA, Pellegrini CA, Wang X, West DS. Describing Transitions in Adherence to Physical Activity Self-monitoring and Goal Attainment in an Online Behavioral Weight Loss Program: Secondary Analysis of a Randomized Controlled Trial. J Med Internet Res. 2022 Jan 28;24(1):e30673. doi: 10.2196/30673. PMID 35089159
- [Derived] West DS, Krukowski RA, Monroe CM, Stansbury ML, Carpenter CA, Finkelstein EA, Naud S, Ogden D, Harvey JR. Randomized controlled trial of financial incentives during weight-loss induction and maintenance in online group weight control. Obesity (Silver Spring). 2022 Jan;30(1):106-116. doi: 10.1002/oby.23322. PMID 34932889
- [Derived] West DS, Krukowski RA, Finkelstein EA, Stansbury ML, Ogden DE, Monroe CM, Carpenter CA, Naud S, Harvey JR. Adding Financial Incentives to Online Group-Based Behavioral Weight Control: An RCT. Am J Prev Med. 2020 Aug;59(2):237-246. doi: 10.1016/j.amepre.2020.03.015. Epub 2020 May 21. PMID 32446752

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Internet Only | Internet + Incentives
Started | 212 | 206
Completed | 172 | 188
Not Completed | 40 | 18
Not completed — Pregnancy | 1 | 3
Not completed — Lost to Follow-up | 38 | 15
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Internet Only | Internet + Incentives | Total
Number analyzed (Participants) | 212 | 206 | 418
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (11.14) | 50 (11.01) | 49 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 187 | 381
  Male | 18 | 19 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 210 | 202 | 412
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 63 | 44 | 107
  White | 147 | 160 | 307
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 212 | 206 | 418
Weight [Mean (Standard Deviation); unit: kilograms] | 97.8 (19.5) | 95.6 (15.9) | 96.7 (17.7)

OUTCOME MEASURES:

1. Primary Outcome: Weight Change
Description: Weight will be measured at baseline, 2, 6 months. Weight loss at 6 months will be calculated as kg lost from baseline.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Internet Only | Internet + Incentives
Number analyzed (Participants) | 212 | 206
kilograms
  Baseline | 97.8 (19.5) | 95.6 (15.9)
  6 Months | 4.7 (6.6) | 6.4 (5.5)
Statistical Analysis 1: Comparison: Internet Only vs Internet + Incentives; The study was designed to detect a 2.2-kg group weight loss difference between groups with a standard deviation of 5.8 kg,4,5 a 5% Type I error rate, and 80% power. To adjust for possible clustering effects in this nested design, the adjusted variance estimate was increased to 7.67, calculated using a conservative intraclass correlation coefficient of 0.05; Test type: Superiority; p < .01, Mixed Models Analysis

2. Secondary Outcome: Class Attendance
Description: Average number of classes attended
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Number of classes attended
Groups:
- Internet Only: Participants will be required to attend a weekly Internet chat session with your group members and one of the behavioral weight control therapists. Participants will learn the principles of managing eating and exercise behaviors in weekly, hour-long chat sessions and by completing weekly lessons. Participants are asked to self-monitor foods and exercise through the use of a smartphone ap. Participants will wear a tracking device that monitors steps. All participants will be contacted via e-mail individually, by their group leader who will monitor their progress and offer advice and encouragement. Meetings are weekly for 24 weeks.
- Internet + Incentives: Participants are given the same intervention as described for the internet only group, with the exception that they will have the opportunity to earn financial incentives. Financial incentives will be based on participants weight loss, and compliance with certain weight loss behaviors including meeting exercise goals, self-monitoring foods consumed, and daily weighing and reporting.
  Internet + Incentives: 6 month behavioral weight loss intervention delivered online with the possibility of earning incentives for losing weight and performing weight loss behaviors including monitoring food intake, exercising, and daily weighing
Arm/Group | Internet Only | Internet + Incentives
Number analyzed (Participants) | 212 | 206
Number of classes attended | 16 (6.6) | 18 (5.1)

3. Secondary Outcome: Self Monitoring of Body Weight
Description: Number of days with body weight self reported
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Number of days weight self report
Groups:
- Internet Only: Participants will be required to attend a weekly Internet chat session with your group members and one of the behavioral weight control therapists. Participants will learn the principles of managing eating and exercise behaviors in weekly, hour-long chat sessions and by completing weekly lessons. Participants are asked to self-monitor foods and exercise through the use of a smartphone app. Participants will wear a tracking device that monitors steps. All participants will be contacted via e-mail individually, by their group leader who will monitor their progress and offer advice and encouragement. Meetings are weekly for 24 weeks.
Arm/Group | Internet Only | Internet + Incentives
Number analyzed (Participants) | 212 | 206
Number of days weight self report | 72 (51) | 115 (43)

4. Secondary Outcome: Dietary Intake Self Monitoring
Description: Number of days reported dietary intake over 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Number of days dietary intake reported
Arm/Group | Internet Only | Internet + Incentives
Number analyzed (Participants) | 212 | 206
Number of days dietary intake reported | 85 (54) | 119 (44)

5. Secondary Outcome: Self Monitoring of Physical Activity
Description: Number of days physical activity reported
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Number of days Physical Activity report
Arm/Group | Internet Only | Internet + Incentives
Number analyzed (Participants) | 212 | 206
Number of days Physical Activity report | 85 (54) | 118 (44)

6. Secondary Outcome: Steps/Day
Description: Number of Steps/day
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: number of steps
Arm/Group | Internet Only | Internet + Incentives
Number analyzed (Participants) | 212 | 206
number of steps | 7447 (2888) | 8057 (2672)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline through 6 months. There were no adverse or serious adverse events to report.
Groups:
- Internet Only: Participants will be required to attend a weekly Internet chat session with your group members and one of the behavioral weight control therapists. Participants will learn the principles of managing eating and exercise behaviors in weekly, hour-long chat sessions and by completing weekly lessons. Participants are asked to self-monitor foods and exercise through the use of a smartphone ap. Participants will wear a tracking device that monitors steps. All participants will be contacted via e-mail individually, by their group leader who will monitor their progress and offer advice and encouragement. Meetings are weekly for 24 weeks and monthly for 12 months.
  Internet Only: 6 month behavioral weight loss intervention delivered online
Arm/Group | Internet Only | Internet + Incentives
All-Cause Mortality (participants affected / at risk) | 0/212 | 0/206
Serious Adverse Events (participants affected / at risk) | 0/212 | 0/206
Other Adverse Events (participants affected / at risk) | 0/212 | 0/206

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-02-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT02688621/Prot_SAP_001.pdf
  • Informed Consent Form (2015-12-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT02688621/ICF_000.pdf